CLINICAL TRIAL: NCT06865742
Title: Effects of Music Therapy Applied During Hemodialysis on Fatigue, Sleep Quality and Mental Well-Being
Brief Title: Music Therapy Applied During Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-mçy
Record Dates: First submitted 2025-02-12; First posted 2025-03-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Music Therapy; Fatigue; Sleep Quality; Mental Well-Being; nursing
MeSH Terms: conditions — Fatigue; Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental type.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music therapy/Experimental group (Experimental): This group will receive music therapy for 30 minutes after the 2nd hour of each hemodialysis session for 4 weeks.
  Interventions: Behavioral: Music intervention
- Control group (No Intervention): No intervention will be performed in this group. Individuals will receive their routine care.

INTERVENTIONS:
Behavioral: Music intervention — This is the first study to evaluate the effects of music therapy on fatigue, sleep quality and mental well-being of individuals receiving HD treatment.
  Arms: Music therapy/Experimental group

SUMMARY:
Many symptoms are encountered during the hemodialysis treatment process, and fatigue and insomnia are two of the most common symptoms. The management of these symptoms, which negatively affect the quality of life and mental well-being of individuals, is very important. It is known that the effects of pharmacological treatments are limited in the management of symptoms encountered during the HD treatment process, and the tendency towards non-pharmacological methods in symptom management is increasing.

This study will be conducted to determine the effects of music therapy to be applied to individuals receiving HD treatment on fatigue, sleep quality and mental well-being.

This randomized controlled experimental study will be conducted with 60 individuals receiving treatment in the hemodialysis clinic of a public hospital. Individuals will receive 30 minutes of music therapy after the 2nd hour of each hemodialysis session for 4 weeks. Research data will be collected using the Introductory Information Form, Chalder Fatigue Scale, Pittsburgh Sleep Quality Scale and Warwick-Edinburgh Mental Well-Being Scale.

This study is important because it is the first study to evaluate the effects of music therapy on fatigue, sleep quality and mental well-being of individuals receiving HD treatment. It is thought that music therapy applied to individuals receiving HD treatment will contribute to the literature on evidence.

DETAILED DESCRIPTION:
Chronic renal failure (CKD) is a disease characterized by progressive and irreversible nephron loss that develops due to various diseases. In the CKD picture, permanent disorders are observed in the fluid-electrolyte balance and metabolic-endocrine functions of the kidney. Although CKD is a disease that can be prevented and/or its progression rate can be slowed down in the early stages, the low level of awareness about the disease and early diagnosis cause the disease to progress to the final stage, end-stage renal failure (ESRD).

Renal replacement therapies (RRT) such as dialysis and kidney transplantation are applied to individuals diagnosed with ESRD. Hemodialysis (HD) is the most commonly used RRT. The aim of HD treatment is to increase the life span and quality of life of individuals. However, it is known that HD, which is one of the life-preserving treatments, causes many undesirable problems in the physical, psychological, social and economic areas in addition to its targeted effects. Individuals who undergo HD encounter many problems such as diet and fluid restriction, job loss, early retirement, role changes and role losses, disruption in family life, dependence on devices and healthcare institutions, fear of death, depression, physical dysfunction, sexual dysfunction, decreased quality of life, and deterioration in body image and self-esteem. In addition, individuals during the treatment process; They also experience many symptoms such as fatigue, shortness of breath, pain, nausea-vomiting, loss of appetite, muscle cramps, insomnia, itching, drowsiness, irritability, dry skin, dizziness, and restlessness.

Fatigue and insomnia are two of the most common symptoms encountered during the HD treatment process. Fatigue, defined as an uncontrollable feeling of exhaustion, is intensely experienced by individuals receiving HD treatment. In the study by Hindistan and Deniz (2018), fatigue was detected in 83.5% of individuals, in the study by Usta and Demir (2014), in 52.2% of individuals before HD, 43.3% during HD, and 84.4% after HD, and in the study by Ju A et al. (2020), in 60-97% of individuals. It is known that fatigue in individuals receiving HD treatment causes an increase in the level of addiction, a decrease in physical activity level, and quality of life. Another problem that causes a decrease in quality of life and also increases the mortality rate is sleep problems. It has been reported that 60-85% of individuals receiving HD treatment have sleep problems. In the study of Taylan and Özkan (2020), it was determined that the sleep quality of individuals receiving HD treatment was low and 41.2% of the individuals had very poor sleep quality. Sleep problems include problems such as prolonged time to fall asleep, interruptions during sleep, daytime naps and restless leg syndrome.

All problems and symptoms encountered during the HD treatment process negatively affect the quality of life and mental well-being of individuals.The management of symptoms experienced in individuals receiving HD treatment is very important due to their effects on the quality of life and mental well-being. It is known that the effects of pharmacological treatments are limited in the management of symptoms encountered during the HD treatment process. Therefore, the tendency towards non-pharmacological methods in the management of these symptoms is increasing. Reducing symptoms in HD and ensuring the well-being of patients has an important place in terms of quality nursing care. For this reason, nurses can take a holistic approach to individuals receiving HD treatment and perform various interventions.In this context, nurses mostly prefer complementary treatments such as massage, aromatherapy, acupuncture, reflexology, and music therapy from non-pharmacological methods.

Music therapy is one of the important complementary treatments preferred by nurses and is a method used to provide symptom management and has no side effects.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being on HD treatment for at least 6 months
* Being cooperative and having no verbal communication disabilities (hearing or speaking)
* Not having a psychiatric disorder

Exclusion Criteria:

* Having recently attended a similar program
* Not agreeing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Is music therapy effective in reducing fatigue? | Baseline and week 4
  The scale is a 4-point Likert type. The physical fatigue subscale score and the mental fatigue subscale score of the scale are added to obtain the general fatigue score. The physical fatigue subscale score can vary between 0-21, the mental fatigue subscale score between 0-12, and the total fatigue score between 0-33. An increase in the scale score indicates an increase in fatigue severity.
Is music therapy effective in improving sleep quality? | Baseline and week 4
  The scale evaluates sleep quality in the last month. It consists of 19 questions and seven subscales, and 18 items are included in the scoring. Each item is evaluated on a 0-3 scale, and the total scale score is the sum of the seven subscale scores. The total score that can be obtained from the scale varies between 0-21, with a high score indicating poor sleep quality. A total scale score of ≤5 indicates "good sleep", and a score of >5 indicates "bad sleep".
Is music therapy effective in improving mental well-being? | Baseline and week 4
  The scale consists of 14 items and is a 5-point Likert type. Scores range from 14 to 70. High scores indicate high psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Karasu, RA, Study Chair — Erzurum Technical University

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.